CLINICAL TRIAL: NCT00596076
Title: The Efficacy of Back School on Low Back Pain and Quality of Life of Workers of a Pharmaceutics Company in Tehran Suburb. COPCORD Study (Stage II)
Brief Title: Back School Efficacy on Low Back Pain and Quality of Life of Workers. COPCORD STUDY (Stage II)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Dr Fereidoon Davatchi, Rheumatology Research Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 85-04-41-4972
Record Dates: First submitted 2008-01-05; First posted 2008-01-16 (Estimated); Last update posted 2010-08-16 (Estimated); Status verified 2010-08

CONDITIONS: Low Back Pain
Keywords: Low back pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Workers with low back pain
  Interventions: Behavioral: Back School

INTERVENTIONS:
Behavioral: Back School — All the workers undergo a clinical examination for low back pain, by two trained practitioner. Those workers who are diagnosed for mechanical low back pain during the last six months fulfill a self report Quality of Life Questionnaire (SF36). The objective level of low back pain will obtain by a visual analogue scale. Then a back school training course will be held in 6 sessions, in 6 consecutive weeks. Two previously trained physiotherapists are responsible for the training course. Each series will have 10 participants. They will learn vertebral column anatomy and its function at the first session. The proper posture and exercises to reduce or inhibit low back pain are taught in the next 4 sessions. The 6th session is arranged for answering questions and checking how exercises are performed.
  A visual analogue scale and quality of life assessment will be held at the end of the last session and the end of the sixth month.

SUMMARY:
The study is an intervention, Phase II COPCORD study. (COPCORD= Community Oriented Program to Control Rheumatic Diseases). The purpose of this study is to find if Back School training has any benefit on low back pain of the workers in a pharmaceutical factory in Tehran suburbs.

DETAILED DESCRIPTION:
A back school will be held on at the Modava Pharmaceutical Factory, in Tehran suburbs. We estimate that this prospective study will include almost one third of the 70 workers in the factory. The study provides objective data and subjective information from patients. The clinical benefits of back school on low back pain and quality of life will be reported at the beginning and the end of intervention and after a period of 6 months follow up.

ELIGIBILITY:
Inclusion Criteria:

* History of mechanical low back pain in the last six months

Exclusion Criteria:

* History of inflammatory spinal diseases
* Severe scoliosis
* History of spinal surgery
* History of spinal malignancy

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2008-02; Primary Completion 2008-03 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
1- Comparison of quality of life in patients with low back pain before and after Back school training. 2- Comparison of low back pain based on a visual analogue scale before and after back school training. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Fereydoun Davatchi, MD, Study Chair — Rheumatology Research Center, Medical Sciences/University of Tehran
Locations (1):
- Rheumatology Research Center, Tehran, Tehran Province, Iran